CLINICAL TRIAL: NCT01484444
Title: Biomarker Analysis of Gastrointestinal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Ki Kang, Professor of Medicine, Sungkyunkwan University School of Medicine, Department of Hematology and Oncology, Samsung Medical Center
Other Study IDs: 2011-07-089
Record Dates: First submitted 2011-11-22; First posted 2011-12-02 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- gastrointestinal cancer

SUMMARY:
BIOMARKER ANALYSES

1. FNA Sample:

   From each enrolled patient who meets the inclusion criteria, FNA sample will only be taken .

   FNA will be carried out only in patients with feasible biopsy or FNA site. Ascites or pleural fluid will be collected for analysis
2. Blood Samples From each enrolled patient who meets the inclusion criteria, blood samples will be collected. 3 mL blood sample will be collected .
3. tumor tissue Archived Tumor Tissue (Slides) Samples Primary tumor and/or a metastatic lesion collected. Approximately 5 unstained slides (if available) are collected.

DETAILED DESCRIPTION:
Recently, a great leap has been accomplished in discovering somatic mutations in human cancer genomes. With the advent of molecularly targeted therapy, somatic mutations have attracted more attention from cancer researchers. Driver mutations confer growth advantage on the cell in which they occur, are causally implicated in cancer development and have therefore been positively selected. In contrast, passenger mutations are biologically neutral and do not confer growth advantage. Hence, driver somatic mutations are conventionally the optimal target for cancer cells. Given the growing evidence of ethnic difference in distribution of somatic mutations, we aim to survey actionable somatic mutations in Asian prevalent cancer.

Ability to assess multiple biomarkers using FNA samples could provide a breakthrough in gastrointestinal cancer clinical studies. FNAs are minimally invasive and, therefore, more acceptable for serial tumor sampling. Furthermore, the cells removed with this method frequently represent relatively pure tumor cell population, and can be processed within minutes after removal from the tumor; therefore, proteomic profiles of FNA specimens likely resemble the in vivo profiles very closely. In addition, tumor cells from metastatic sites obtained using FNA may provide site specific metastatic tumor profile. Acquired resistances to therapies is well known in various cancer types.1, 2 Serial sampling of tumor tissue by FNA will provide important resources to monitor tumor changes as a function of time and therapy.

There have been numerous studies reporting the detection of carcinoma cells in the blood of patients with solid tumors. Detection of CTCs (Circulating Tumor Cells) before initiation of first-line therapy in patients with metastatic breast cancer is highly predictive of progression free survival and overall survival.3-5 These studies led to the FDA clearance of the vertex CellSearch technology. The prognostic implication of detecting CTCs prior to initiating therapy raises important questions about the biological attributes of these cells. CTCs are found in most metastatic diseases and it may be reflective of the status of the recurrent tumor looking for alternate site to colonize. However, not all CTCs would successfully establish metastatic colonies. Having the ability to profile tumors at different metastatic sites together with CTCs could provide information on the subset of most robust CTCs with highest metastatic potentials. In addition CTCs could provide alternative source of tumor cells that may be used to detect tumor changes as the cancer progresses and therapy continued or modified.

The expression/activation profiling of kinases and other signal transduction pathway molecules along with markers critical for triggering angiogenesis on a serial sampling of tumor and tumor associated tissues will provide valuable information on changes occurring in tumor cells as a function of time and therapies. This temporal and spatial profiling of tumor progression will enable clinicians to monitor rapidly 'evolving' cancer signatures in each patient. The temporal and site-specific profiling of CTCs and FNAs must then utilize highly sensitive and specific method to interrogate limited amount of cancer cells in such samples. Based on these results, we plan to design genome-directed clinical trials in these tumor types.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed gastrointestinal cancer.
* Patients should sign a written informed consent .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastrointestinal cancer Patients.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Analyzed of DNA mutations | 24months
  To estimate genotypes concerning DNA repair (ERCC1, XPD, XRCC1) and detoxification (GSTP1)

CONTACTS AND LOCATIONS:
Overall Officials: won ki kang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung medical Center, Seoul, South Korea